CLINICAL TRIAL: NCT03610464
Title: Pharmacokinetic Study of DYANAVEL XR (Amphetamine) Extended-release Oral Suspension, in Children Aged 4 to 5 Years With Attention-deficit/Hyperactivity Disorder
Brief Title: Pharmacokinetic Study of DYANAVEL XR (Amphetamine) Extended-release Oral Suspension, in Children Aged 4 to 5 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRI102-PPK-300
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Intervention Model Description: This was an open-label, single-site, single-dose one-period, one-treatment study in 5 pediatric subjects diagnosed with ADHD, otherwise healthy. Subjects received a single, 1 mL dose of AMPH EROS 2.5 mg/mL, from which PK was assessed over a 28 hour period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study patients (AMPH EROS) (Experimental): All patients treated with extended-release oral suspension (AMPH EROS) that contains 2.5 mg/mL amphetamine base
  Interventions: Drug: Amphetamine Extended Release Suspension [Dyanavel]

INTERVENTIONS:
Drug: Amphetamine Extended Release Suspension [Dyanavel] — 1 mL of study drug (AMPH EROS, 2.5 mg/mL), pharmacokinetic analysis
  Other Names: DYANAVEL XR, amphetamine extended release oral suspension

SUMMARY:
The objective of this study was to evaluate the plasma amphetamine concentration/time profile of amphetamine extended release oral suspension in children aged 4 to 5 years with attention-deficit/hyperactivity disorder, following a single 2.5 mg dose of amphetamine extended release oral suspension.

DETAILED DESCRIPTION:
DYANAVEL® XR is an extended-release oral suspension that contains 2.5 mg/mL amphetamine base (amphetamine extended-release oral suspension; AMPH EROS). Drug-resin complexation is formed with the amphetamine and sodium polystyrene sulfonate, an ion exchange resin. The extended release feature of the product is achieved by coating a portion of the drug/resin complexes with an extended release coating. AMPH EROS contains approximately a 3.2:1 ratio of d-amphetamine compared to l-amphetamine.

The objective of this study was to evaluate the plasma amphetamine concentration/time profile of AMPH EROS in children aged 4 to 5 years with attention-deficit/hyperactivity disorder, following a single 2.5 mg dose of AMPH EROS.

These data will guide appropriate dosing in planned safety and efficacy studies with AMPH EROS in a preschool population with attention-deficit/hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 4 to 5 years at the time of enrollment into this study;
2. Body weight ≥ 28 lb. at screening visit;
3. Diagnosed with ADHD by a psychiatrist, psychologist, developmental pediatrician, pediatrician, or an experienced licensed allied health professional approved by the Sponsor by using the DSM-5 criteria and supported by a structured Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL) interview, administered at the Screening Visit (Visit 0);
4. Provide written informed consent (parent/guardian) prior to participation in the study.

Exclusion Criteria:

1. Diagnosed with any DSM-5 active disorder (other than ADHD) with the exception of specific phobias, learning disorders, motor skills disorders, communication disorders,oppositional defiant disorder, elimination disorders, and sleep disorders
2. History of chronic medical illnesses including seizure disorder (excluding a history of febrile seizures), moderate to severe hypertension, untreated thyroid disease, known structural cardiac disorders, serious cardiac conditions, serious arrhythmias, cardiomyopathy and known family history of sudden death
3. Known history or presence of significant renal or hepatic disease, as indicated by clinical laboratory assessment (liver function test results ≥ 2 times the upper limit of normal, blood urea nitrogen, or creatinine)
4. Clinically significant (CS) abnormal ECG or cardiac findings on physical examination (including the presence of a pathologic murmur)
5. Use of the following medications within 30 days of dosing:

   * MAOI - monoamine oxidase inhibitors (e.g., Selegiline, isocarboxazid, phenelzine, tranylcypromine);
   * Tricyclic Antidepressants (e.g. Desipramine, protriptyline);
6. Use of the following medications within 3 days of dosing

   * Gastrointestinal acidifying agents (e.g., guanethidine, reserpine, glutamic acid HCl, ascorbic acid);
   * Urinary acidifying agents (e.g., ammonium chloride, sodium acid phosphate,methenamine salts);
7. Use of atomoxetine within 14 days of dosing
8. Planned use of prohibited drugs or agents from the screening visit through the end of the study. Medications used to support sleep may be acceptable with the written approval of the sponsor or medical monitor
9. Abnormal CS laboratory test value at screening that, in the opinion of the sponsor or medical monitor, would preclude study participation
10. Known history of allergy/hypersensitivity to amphetamine or any of the components of AMPH EROS, heparin flush and topical anesthetics
11. Parent or guardian's inability or unwillingness to follow directions of the Investigator or study research staff
12. Any uncontrolled medical condition that in the opinion of the Investigator would preclude study participation
13. History of significant illness requiring hospitalization, or surgery requiring anesthetics within 30 days of dosing.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pardo, MD, Study Director — Tris Pharma, Inc.
Locations (1):
- Meridien Research, Inc., Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Patients (AMPH EROS)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat
Arm/Group | Study Patients (AMPH EROS)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 16.2 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentrations of d- and L-amphetamine
Description: Plasma Concentration of d- and l-amphetamine measured at 0, 1, 3, 4, 6, 8, 10, 12, and 28 hours postdose.
Time Frame: 0-28 hours postdose
Population: intention to treat population
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Plasma Concentration of d-Amphetamine; Plasma Concentration of l-Amphetamine: All patients treated with extended-release oral suspension (AMPH EROS) that contains 2.5 mg/mL amphetamine base
  Amphetamine Extended Release Suspension [Dyanavel]: 1 mL of study drug (AMPH EROS, 2.5 mg/mL), pharmacokinetic analysis
Arm/Group | Plasma Concentration of d-Amphetamine | Plasma Concentration of l-Amphetamine
Number analyzed (Participants) | 5 | 5
ng/mL
  0 hours postdose | 0 (0) | 0 (0)
  1 hour postdose | 3.5 (3.0) | 1.1 (0.9)
  3 hours postdose | 19.9 (2.2) | 6.2 (0.7)
  4 hours postdose | 20.2 (2.5) | 6.4 (0.8)
  6 hours postdose | 17.5 (3.2) | 5.7 (1.1)
  8 hours postdose | 16.9 (2.2) | 5.6 (0.8)
  10 hours postdose | 14.4 (3.3) | 4.8 (1.1)
  12 hours postdose | 11.6 (3.2) | 3.9 (1.1)
  28 hours postdose | 2.2 (0.7) | 0.9 (0.2)

ADVERSE EVENTS:
Time Frame: 48 hours post-dose. Pharmacokinetics study.
Arm/Group | Study Patients (AMPH EROS)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03610464/Prot_SAP_000.pdf